CLINICAL TRIAL: NCT07081490
Title: The Effect of Training Provided With Virtual Escape Room Game on Nurses' Knowledge Level on Pressure Injury Regarding Medical Devices
Brief Title: Virtual Escape Room Game About Medical Device in Nurses
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kahramanmaraş İstiklal University (Other)
Responsible Party: Principal Investigator, Nurhan Aktaş, assistant professor, Kahramanmaraş İstiklal University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: KIstiklal University
Record Dates: First submitted 2025-07-11; First posted 2025-07-23 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Nursing Caries; Pressure Injuries
Keywords: Escape room; Gamification; Digital game; Pressure Injuries
MeSH Terms: conditions — Pressure Ulcer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- virtual escape room game group (Experimental): A virtual escape room gaming group is a group that plays a virtual escape room game. Virtual escape rooms are remotely accessible digital versions of physical escape rooms. Virtual escape rooms are adaptations of physical escape rooms that use online interactive environments where participants aim to solve puzzles within a set timeframe.
  Interventions: Other: Virtual Escape Room Game

INTERVENTIONS:
Other: Virtual Escape Room Game — Virtual escape rooms are digital versions of physical escape rooms that can be accessed remotely. Virtual escape rooms are adaptations of physical escape rooms that use online interactive environments where participants aim to solve puzzles within a set timeframe.

SUMMARY:
The research was planned as a pre-test-post-test single-group, quasi-experimental design in order to develop a web-based digital education game to improve nurses' knowledge level on pressure injuries related to medical devices and to evaluate the effect of the developed game on nurses' knowledge acquisition on pressure injuries related to medical devices, as well as the use of the game and user experience. The sample of the research will consist of nurses working in the intensive care unit at Kahramanmaraş Necip Fazıl City Hospital who meet the research criteria and agree to participate in the research. In the first stage of the research, the materials necessary for the game development and evaluation process will be prepared and the content validity study of these materials will be conducted. In the second stage, the development and preliminary evaluation of the virtual escape room game will be done. In the third stage, the virtual escape room game will be applied and data will be collected. Data will be collected from the nurses with the 'Introductory Features Form' and the 'Medical Device Related Pressure Injury Knowledge Level Assessment Test' (pre-test) before the game application; and after the game application, the 'Medical Device Related Pressure Injury Knowledge Level Assessment Test' (post-test) and the Virtual Escape Room Game Evaluation Form. After 4 weeks of the game application (retest), nurses will be asked to answer the questions of the 'Medical Device-Related Pressure Injury Knowledge Level Assessment Test'.

H1a: What is the effect of the virtual escape room game on nurses' knowledge levels regarding TCBBY? H1b: What are the usage and user experiences of the virtual escape room game developed for the purpose of educating nurses on the prevention of TCBBY?

DETAILED DESCRIPTION:
The research was planned as a pre-test-post-test, single-group, quasi-experimental design in order to develop a web-based digital education game to improve nurses' knowledge level about pressure injuries related to medical devices and to evaluate the effects of the developed game on nurses' knowledge acquisition about pressure injuries related to medical devices, the use of the game, and the user experience. The universe of the research will consist of nurses working in the intensive care unit of Kahramanmaraş State Hospital. It is planned to reach the universe in the research and no sample calculation has been made. The sample of the research will consist of nurses working in the intensive care unit of Kahramanmaraş Necip Fazıl City Hospital who meet the research criteria and agree to participate in the research. In the first stage of the research, the materials necessary for the game development and evaluation process will be prepared and the content validity study of these materials will be conducted. In the second stage, the development and preliminary evaluation of the virtual escape room game will be done. In the third stage, the virtual escape room game will be applied and data will be collected. The data will be collected by filling out the 'Introductory Characteristics Form' and 'Medical Device Related Pressure Injury Knowledge Level Assessment Test' (pre-test) to the nurses before the game application; After the game application, the data will be collected with the 'Medical Device Related Pressure Injury Knowledge Level Assessment Test' (post-test) and the Virtual Escape Room Game Evaluation Form. After 4 weeks of the game application (re-test), the nurses will be asked to answer the 'Medical Device Related Pressure Injury Knowledge Level Assessment Test' questions. The analysis of the data will be completed by transferring it to the IBM SPSS Statistics 23 program. Frequency distribution (number, percentage) will be given for categorical variables, and descriptive statistics (mean, standard deviation, minimum, maximum) will be given for numerical variables. Parametric and non-parametric tests will be used according to the normal distribution of the data.

ELIGIBILITY:
Inclusion Criteria:

* Volunteering to participate in the study
* Working as a nurse in an intensive care unit at the time of the study
* Having internet access
* Being able to use a computer

Exclusion Criteria:

* Not completing data collection forms or providing incomplete answers.
* Having received any prior training on medical device-related pressure injuries.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-07-20 (Estimated); Primary Completion 2025-09-20 (Estimated); Study Completion 2025-12-20 (Estimated)

PRIMARY OUTCOMES:
Nurses' knowledge level regarding medical device-related pressure injuries | Before the virtual escape room game
  The Medical Device-Associated Pressure Injury Knowledge Level Assessment Test (MDAPIKLAT) is administered to nurses.
  It is a multiple-choice test developed by Dalli and Girgin (2023) to assess nurses' knowledge of pressure injuries related to medical devices and has undergone psychometric validation. The test consists of 16 questions covering six themes (Theme 1: Diagnosis and Etiology, Theme 2: Staging and Observation, Theme 3: Medical Device Selection and Suitability, Theme 4: Skin Assessment, Theme 5: Prevention, Theme 6: Special Patient Groups) related to pressure injuries associated with medical devices. Correct answers are scored as 1, incorrect or blank answers are scored as 0. The total score ranges from 0 to 16. The item difficulty index of the questions was found to be 0.36-0.84, and the item discrimination values were found to be 0.31-0.68. The correlation coefficient of the test was 0.82, and the overall internal consistency reliability was 0.77.

SECONDARY OUTCOMES:
Knowledge level of nurses regarding medical device-related pressure injuries after the virtual escape room game | one week after the virtual escape room game
  After the virtual escape room game, the knowledge level of the nurses is evaluated with the Medical Device Associated Pressure Injury Knowledge Level Assessment Test (MDAPIKLAT).
  MDAPIKLAT: multiple-choice test was developed by Dalli and Girgin (2023) to assess nurses' knowledge of pressure injuries related to medical devices and has undergone psychometric validation. The test consists of 16 questions covering six themes (Theme 1: Diagnosis and Etiology, Theme 2: Staging and Observation, Theme 3: Medical Device Selection and Suitability, Theme 4: Skin Assessment, Theme 5: Prevention, Theme 6: Special Patient Groups) related to pressure injuries related to medical devices. Correct answers are scored as 1, incorrect or blank answers are scored as 0. The total score ranges from 0 to 16. The item difficulty index of the test questions was found to be 0.36-0.84, and the item discrimination values were found to be 0.31-0.68.
Nurses' perception of virtual escape room game experience | one week after the virtual escape room game
  Nurses' post-virtual escape room game experiences are evaluated with the Gameful Experience Scale (GAMEX).
  GAMEX:The scale, developed by Eppman et al. (2018), and whose validity and reliability study in Turkish was conducted with nursing students by Çömez İkican et al. (2024), is used to assess game experience. The scale consists of a total of 27 items and 5 subdimensions. The subdimensions are enjoyment, immersion in play, creative thinking and emotional activation, absence of negative effects, and mastery. A 5-point Likert-type scale is used in the evaluation of the scale, with scores of "Never" (1), "Rarely" (2), "Occasionally" (3), "Frequently" (4), and "Always" (5). Items 18, 21, 22, and 23 of the scale are scored reversely ("Never" (5), "Rarely" (4), "Occasionally" (3), "Frequently" (2), and "Always" (1). In the original and validity-reliability study of the scale, the Cronbach alpha value for the entire scale was found to be 0.89.

CONTACTS AND LOCATIONS:
Locations (1):
- Kahramanmaraş Istiklal University, Kahramanmaraş, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No